CLINICAL TRIAL: NCT00306124
Title: Dopaminergic Enhancement of Learning and Memory (LL_001, Project on Dementia/MCI)
Brief Title: Dopaminergic Enhancement of Learning and Memory in Healthy Adults and Patients With Dementia/Mild Cognitive Impairment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LL_001 Project on Dementia/MCI
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2007-10-25 (Estimated); Status verified 2007-10

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment; Healthy
Keywords: Dementia; Mild Cognitive Impairment; MCI; levodopa; learning; enhancement
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia | interventions — Levodopa

INTERVENTIONS:
Drug: Levodopa

SUMMARY:
This study aims to determine whether levodopa is effective in boosting learning and memory in healthy subjects and patients with dementia or Mild Cognitive Impairment.

We also examine in healthy subjects using functional magnetic resonance imaging which brain regions mediate improved learning after levodopa administration.

DETAILED DESCRIPTION:
Prior work of our group shows that the dopamine precursor levodopa markedly improves word learning success in healthy subjects. In this randomized, placebo-controlled, double-blind trial, we probe whether administration of levodopa improves learning performance as compared to placebo administration on neuropsychological tests and in an associative learning paradigm. We postulate that levodopa improves learning success and memory performance in healthy subjects, while the effect in patients with dementia or Mild Cognitive Impairment might depend on other factors, including severity of memory impairment.

ELIGIBILITY:
Inclusion criteria for patients with dementia:

* Patients: clinical diagnosis of AD or mild cognitive impairment
* primary language German

Exclusion Criteria for healthy subjects and patients with dementia/MCI:

* Known allergy to levodopa or tetrazine
* History of medication/drug abuse
* Acute nicotine withdrawal or > 15 cigarettes per day
* > 6 cups/glasses of coffee, caffeine drinks or energy drinks per day
* > 50 grams of alcohol per day
* Severe hypertonia (systole >160 mm Hg)
* Severe arteriosclerosis
* Diabetes, asthma, or glaucoma
* Severe hearing disability
* no focal brain lesions
* Premorbid depression or psychosis
* Medication with dopamine agonists or antagonists
* Parkinsonian symptoms

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-01; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Cognitive performance assessed by neuropsychological tests and learning paradigms under placebo and levodopa in healthy subjects and patients with dementia or Mild Cognitive Impairment.
Brain activity pattern during learning under levodopa as compared to placebo in healthy subjects.

SECONDARY OUTCOMES:
Long-term stability of learning performance after 1 month in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Knecht, MD, Principal Investigator — Neurology, University of Muenster, Germany; Caterina Breitenstein, PhD, Principal Investigator — Neurology, University of Muenster, Germany; Julia Reinholz, PhD, Study Director — Neurology, University of Muenster, Germany
Locations (1):
- University of Muenster, Department of Neurology, Münster, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Knecht S, Breitenstein C, Bushuven S, Wailke S, Kamping S, Floel A, Zwitserlood P, Ringelstein EB. Levodopa: faster and better word learning in normal humans. Ann Neurol. 2004 Jul;56(1):20-6. doi: 10.1002/ana.20125. PMID 15236398
- [Background] Breitenstein C, Knecht S. [Language acquisition and statistical learning]. Nervenarzt. 2003 Feb;74(2):133-43. doi: 10.1007/s00115-002-1466-1. German. PMID 12596014
- [Background] Floel A, Hummel F, Breitenstein C, Knecht S, Cohen LG. Dopaminergic effects on encoding of a motor memory in chronic stroke. Neurology. 2005 Aug 9;65(3):472-4. doi: 10.1212/01.wnl.0000172340.56307.5e. PMID 16087920